CLINICAL TRIAL: NCT05493670
Title: Role of Subthalamic Nucleus in Speech and Movement Among People With Parkinson's Disease as Revealed by Intraoperative Recordings and Deep Brain Stimulation
Brief Title: Subthalamic Nucleus Deep Brain Stimulation in Speech Study
Acronym: SiSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jeremy Greenlee (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Pittsburgh (Other); University at Buffalo (Other); Northwestern University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Jeremy Greenlee, Professor of Neurosurgery, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202001213; R01DC017718 (NIH)
Record Dates: First submitted 2021-04-09; First posted 2022-08-09 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease; Dysarthria
Keywords: Deep Brain Stimulation; Parkinson; Speech; Movement; Intelligibility
MeSH Terms: conditions — Parkinson Disease; Dysarthria; Speech

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DBS-STN: The DBS-STN group will consist of individuals with Parkinson's disease who have already elected to undergo deep brain stimulation surgery.
- Control: The control group will consist of individuals with Parkinson's disease who are not undergoing deep brain stimulation placement. No interventions will be completed with the control group.

SUMMARY:
Parkinson's disease (PD) patients treated with deep brain stimulation (DBS) of the subthalamic nucleus (STN) have unpredictable and varied speech outcomes after this treatment. Our research will prospectively document speech performance before, during and 6- and 12-months after STN-DBS in 80 surgically treated patients and compared with 40 non-surgical controls with Parkinson's disease. This study will provide unique insights into the role of STN in speech production, document speech outcome in a comprehensive fashion, identify factors that predict functional communication ability 12 months after STN-DBS, and test the feasibility of low frequency DBS in reversing DBS-induced speech declines in order to optimize treatment strategies for those living with Parkinson's disease.

DETAILED DESCRIPTION:
Aim 1. Define the mechanistic role of STN in speech using direct intraoperative brain recordings. For the first time, we will define STN neuronal physiology for both speech and limb tasks. Through multichannel microelectrode recording (MER) during awake STN-DBS implantation surgery, we will test the hypothesis suggested by our pilot data that STN firing rate during speech will be significantly different from the firing rate during a limb motor task.

Aim 2. Advance understanding of speech outcomes associated with STN-DBS. Intelligibility will serve as the primary functional communication outcome, with communication participation as a secondary metric. Acoustic measures of articulation, phonatory-respiratory behavior and tempo-fluency will be obtained.

Aim 2A. Determine differential effects of DBS stimulation (ON vs. OFF) on speech outcomes. ON vs. OFF stimulation changes in acoustic measures of speech will be used to inform potential reasons for observed changes in intelligibility.

Aim 2B. Define longitudinal effects of STN-DBS on speech outcomes. Speech outcomes and limb measures obtained pre-surgery will be compared to those at 6 and 12 months post-surgery when DBS stimulation is ON. Change in communication participation also will be defined. The control group studied at similar time points will control for disease progression.

Aim 2C. Determine associations between acoustic measures and intelligibility in STN-DBS.

Aim 3. Explore factors associated with changes in intelligibility post STN-DBS. As initial endeavors to guide future studies, we will:

Aim 3A. Use our metrics from Aims 1 and 2 (e.g. disease-specific characteristics, microelectrode recording data, pre-operative intelligibility) to identify factors that predict intelligibility at 12 months following STN-DBS.

Aim 3B. Test the feasibility of manipulating DBS stimulation parameters to improve intelligibility in a subset of participants with DBS-induced intelligibility declines.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in this study, participants must

* have a confirmed diagnosis of idiopathic Parkinson's disease and no atypical Parkinsonism features
* experience significant motor fluctuations
* currently taking and responsive to dopaminergic medications (e.g. Levodopa)
* use English as their primary language
* lack significant cognitive impairment and be able to consent to participate

Exclusion Criteria:

* Significant hearing loss/reliance on hearing aids

Ages: 21 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit 80 STN-DBS participants and 40 participants with Parkinson's disease to serve as non-surgical controls. All Parkinson's disease patients judged to be candidates for DBS surgery by the implanting neurosurgeon and movement disorder neurologists who decide to undergo bilateral surgery will be considered candidates for the study. Control subjects must have a diagnosis of Parkinson's disease and no plan to undergo DBS surgery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Neuron Firing Rate | Intraoperatively
  DBS-STN participants will complete simple speech and motor tasks during surgery while the surgeon records neuron firing rate using Microelectrode Recording (MER).

SECONDARY OUTCOMES:
Speech Intelligibility with DBS ON | Speech intelligibility with DBS ON will be measured at the 6 month follow up and 12 month follow up for the DBS-STN group.
  Speech intelligibility will be measured using the Sentence Intelligibility Test (SIT). Speech intelligibility ratings are measured as percentages, with lower percentages indicating more severe speech impairments.
Speech Intelligibility (stimulation OFF or not applicable) | Speech intelligibility without stimulation will be measured at baseline, 6 month, and 12 month visits for all participants.
  Speech intelligibility will be measured using the Sentence Intelligibility Test (SIT). Speech intelligibility ratings are measured as percentages, with lower percentages indicating more severe speech impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Greenlee, MD, Principal Investigator — University of Iowa Dept of Neurosurgery
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sidtis D, Sidtis JJ. Subcortical Effects on Voice and Fluency in Dysarthria: Observations from Subthalamic Nucleus Stimulation. J Alzheimers Dis Parkinsonism. 2017;7(6):392. doi: 10.4172/2161-0460.1000392. Epub 2017 Oct 30. PMID 29456879
- [Background] Sidtis JJ, Alken AG, Tagliati M, Alterman R, Van Lancker Sidtis D. Subthalamic Stimulation Reduces Vowel Space at the Initiation of Sustained Production: Implications for Articulatory Motor Control in Parkinson's Disease. J Parkinsons Dis. 2016 Mar 19;6(2):361-70. doi: 10.3233/JPD-150739. PMID 27003219
- [Background] Skodda S. Effect of deep brain stimulation on speech performance in Parkinson's disease. Parkinsons Dis. 2012;2012:850596. doi: 10.1155/2012/850596. Epub 2012 Nov 21. PMID 23227426
- [Background] Sturman MM, Vaillancourt DE, Metman LV, Bakay RA, Corcos DM. Effects of five years of chronic STN stimulation on muscle strength and movement speed. Exp Brain Res. 2010 Sep;205(4):435-43. doi: 10.1007/s00221-010-2370-8. Epub 2010 Aug 10. PMID 20697699
- [Background] Tourville JA, Guenther FH. The DIVA model: A neural theory of speech acquisition and production. Lang Cogn Process. 2011 Jan 1;26(7):952-981. doi: 10.1080/01690960903498424. PMID 23667281
- [Background] Dayal V, Limousin P, Foltynie T. Subthalamic Nucleus Deep Brain Stimulation in Parkinson's Disease: The Effect of Varying Stimulation Parameters. J Parkinsons Dis. 2017;7(2):235-245. doi: 10.3233/JPD-171077. PMID 28505983
- [Background] Pal PK, Lee CS, Samii A, Schulzer M, Stoessl AJ, Mak EK, Wudel J, Dobko T, Tsui JK. Alternating two finger tapping with contralateral activation is an objective measure of clinical severity in Parkinson's disease and correlates with PET. Parkinsonism Relat Disord. 2001 Oct;7(4):305-309. doi: 10.1016/s1353-8020(00)00048-1. PMID 11344014
- [Background] Lipski WJ, Alhourani A, Pirnia T, Jones PW, Dastolfo-Hromack C, Helou LB, Crammond DJ, Shaiman S, Dickey MW, Holt LL, Turner RS, Fiez JA, Richardson RM. Subthalamic Nucleus Neurons Differentially Encode Early and Late Aspects of Speech Production. J Neurosci. 2018 Jun 13;38(24):5620-5631. doi: 10.1523/JNEUROSCI.3480-17.2018. Epub 2018 May 22. PMID 29789378
- [Background] Seifried C, Weise L, Hartmann R, Gasser T, Baudrexel S, Szelenyi A, van de Loo S, Steinmetz H, Seifert V, Roeper J, Hilker R. Intraoperative microelectrode recording for the delineation of subthalamic nucleus topography in Parkinson's disease. Brain Stimul. 2012 Jul;5(3):378-387. doi: 10.1016/j.brs.2011.06.002. Epub 2011 Jul 8. PMID 21782543
- [Background] Hebb AO, Darvas F, Miller KJ. Transient and state modulation of beta power in human subthalamic nucleus during speech production and finger movement. Neuroscience. 2012 Jan 27;202:218-33. doi: 10.1016/j.neuroscience.2011.11.072. Epub 2011 Dec 6. PMID 22173017
- [Background] Dromey C, Kumar R, Lang AE, Lozano AM. An investigation of the effects of subthalamic nucleus stimulation on acoustic measures of voice. Mov Disord. 2000 Nov;15(6):1132-8. doi: 10.1002/1531-8257(200011)15:63.0.co;2-o. PMID 11104196